CLINICAL TRIAL: NCT03548922
Title: Impact of Risser Stage on Pressure of Correction in Pectus Carinatum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.327
Record Dates: First submitted 2018-05-20; First posted 2018-06-07 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Pectus Carinatum
Keywords: Risser; Tanner; pressure of correction
MeSH Terms: conditions — Pectus Carinatum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pectus carinatum: Demographic data (age, sex), pressure of correction, Tanner stage, Risser stage, Haller index, pectus carinatum protrusion measurements of patients with pectus carinatum will be recorded and association of them with pressure of correction will be investigated.
  Interventions: Other: Tanner stage; Other: Risser stage; Other: Pressure of correction; Other: Pectus carinatum protrusion

INTERVENTIONS:
Other: Tanner stage — a scale of pubertal development in children, adolescents
Other: Risser stage — a measure showing the growth left in the spine
Other: Pressure of correction — an indirect parameter of the chest wall's flexibility. It is defined as the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax.
Other: Pectus carinatum protrusion — distance from the point of maximum protrusion to the estimated normal level of chest wall

SUMMARY:
Pectus carinatum (PC) is a deformity of the anterior chest wall which is a common pediatric condition, characterized by an idiopathic overgrowth of the costal cartilages resulting in protrusion of the sternum. Knowing factors influencing pressure of correction may lead successful treatment outcomes. In a study by Lee and colleagues investigating the effectiveness of the orthosis, it was found that patients with advanced Tanner stage of pubertal development had a longer time for correction of deformity. Martinez-Ferro et al proposed that pectus carinatum may return mildly, in approximately 10% of cured patients, particularly if they have been treated before pubertal growth spurts or in case they have cured very rapidly. To the best of our knowledge factors influencing pressure of correction and treatment outcomes after compressive bracing have not been investigated before. Our aim is to investigate impact of Risser stage on pressure of correction in PC.

DETAILED DESCRIPTION:
Pectus carinatum (PC) is a deformity of the anterior chest wall which is a common pediatric condition, characterized by an idiopathic overgrowth of the costal cartilages resulting in protrusion of the sternum. Chest pain or discomfort, especially when lying in prone position, increased respiratory effort during exercise, scoliosis, impaired shoulders and kyphotic position are some of the physical signs and symptoms. Unlike pectus excavatum, PC is rarely associated with significant cardiopulmonary involvement except in severe cases. Pectus carinatum is not just a simple aesthetical problem. It can be responsible of physical signs and symptoms and also has significant psychological impact. The classical management of pectus deformities, both carinatum and excavatum, has been primarily surgical. Modification of the Ravitch technique involves resection of the deformed costal cartilages along with sternal osteotomy. Because the results of this technique resulted in worse cosmetic results, a new less invasive procedure, the Nuss procedure was developed. Nuss procedure includes remodeling of the chest wall cartilage with an internal support bar. These techniques have demonstrated the plasticity of the chest wall and led clinicians to hypothesize that carinatum defects would also remodel in response to chronic pressure, leading to a cosmetically superior, nonoperative technique: compression brace. Compression brace is a dynamic orthosis which is custom-fitted, rigid aluminum brace that is adjustable to any thoracic shape. Complications of brace use include uncommon (4.6%), mild and easy to resolve: back pain, hematoma and skin ulceration. Pressure of correction is the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax. It is an indirect parameter of the chest wall's flexibility. It can be measured with a pressure measuring device in pounds per square inches (PSI). Some special designed braces contain a part in which pressure measuring device can be docked. This enables measuring of pressure of treatment. Pressure of treatment can be different from pressure of correction since skin breakdown occurs with corrections at high pressure.

In the Calgary protocol, wearing brace 23 hours a day during the correction phase until the development of the axial skeleton is completed and afterwards 8 hours of wear is recommended in the continuation phase. Marcelo Martinez-Ferro et al developed pressure measuring device and special designed braces contain a part in which pressure measuring device can be docked. They suggested that patients with pressure of correction <10 should be braced. De Beer et al. also recommended the surgical treatment in the presence of chondro-manubrial type PC and pressure of correction > 10 PSI.

Knowing factors influencing pressure of correction may lead successful treatment outcomes. In a study by Lee and colleagues investigating the effectiveness of the orthosis, it was found that patients with advanced Tanner stage of pubertal development had a longer time for correction of deformity. Marcelo Martinez-Ferro et al proposed that pectus carinatum may return mildly, in approximately 10% of cured patients, particularly if they have been treated before pubertal growth spurts or in case they have cured very rapidly.

In general, the long bone growth plates close at 15 to 17 years in males and 13 to 15 years of age in females. An accurate way to determine the skeletal age of a child is to use an X ray of the left wrist and to compare it with X rays in the Greulich and Pyle atlas. Here a series of X rays showing the development and ossification of the wrist, and hand bones is displayed, together with the average age these appear. The axial skeleton matures a few years later than the limbs, and for scoliosis, the Risser sign is a useful method of bone age determination. Skeletal age can be determined by the appearance of the iliac apophysis of the pelvis. The apophysis appears laterally on a pelvic X ray and moves towards the spine as the patient approaches adulthood. Risser's sign is a measure the growth left in the spine - this may help to determine the potential for progression of scoliosis.

To the best of our knowledge factors influencing pressure of correction and treatment outcomes after compressive bracing have not been investigated before. Our aim is to investigate impact of Risser stage on pressure of correction in PC. Demographic data (age, sex), pressure of correction, Tanner stage, Risser stage, Haller index, pectus carinatum protrusion measurements of patients with PC will be recorded and association of them with pressure of correction will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Chondro-gladiolar pectus carinatum (PC)
2. Patients with PC between the ages of 8-24 years

Exclusion Criteria:

1. Patients who previously used compression brace
2. Chondro-manubrial PC
3. Severe scoliosis (Cobb angle>20 degrees)
4. Systemic chronic disease
5. Complex anomaly, PC as a part of syndrome
6. he history of surgical correction of scoliosis or pectus deformity.

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with pectus carinatum who never experienced brace before
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Risser (a measure showing the growth left in the spine) | Day 0
  stage 0: no ossification center at the level of iliac crest apophysis stage 1: apophysis under 25% of the iliac crest stage 2: apophysis over 25-50% of the iliac crest stage 3: apophysis over 50-75% of the iliac crest stage 4: apophysis over >75% of the iliac crest stage 5: complete ossification and fusion of the iliac crest apophysis

SECONDARY OUTCOMES:
Tanner (a scale of physical pubertal development in children, adolescents and adults) | Day 0
  a scale of physical pubertal development in children, adolescents and adults.
pressure of correction (an indirect parameter of the chest wall's flexibility. It is defined as the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax) | Day 0
  an indirect parameter of the chest wall's flexibility. It is defined as the pressure applied to the patient, in the most protruding area of the chest, needed to accomplish a proper shape of the thorax.
Pectus carinatum protrusion (distance from the point of maximum protrusion to the estimated normal level of chest wall) | Day 0
  distance from the point of maximum protrusion to the estimated normal level of chest wall

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Yuksel, Prof, Study Chair — Marmara University; Gulseren Akyuz, Prof, Study Director — Marmara University; Esra Giray, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fokin AA, Steuerwald NM, Ahrens WA, Allen KE. Anatomical, histologic, and genetic characteristics of congenital chest wall deformities. Semin Thorac Cardiovasc Surg. 2009 Spring;21(1):44-57. doi: 10.1053/j.semtcvs.2009.03.001. PMID 19632563
- [Background] Martinez-Ferro M, Bellia Munzon G, Fraire C, Abdenur C, Chinni E, Strappa B, Ardigo L. Non-surgical treatment of pectus carinatum with the FMF(R) Dynamic Compressor System. J Vis Surg. 2016 Mar 17;2:57. doi: 10.21037/jovs.2016.02.20. eCollection 2016. PMID 29078485
- [Background] Kravarusic D, Dicken BJ, Dewar R, Harder J, Poncet P, Schneider M, Sigalet DL. The Calgary protocol for bracing of pectus carinatum: a preliminary report. J Pediatr Surg. 2006 May;41(5):923-6. doi: 10.1016/j.jpedsurg.2006.01.058. PMID 16677884
- [Background] de Beer SA, Gritter M, de Jong JR, van Heurn ELW. The Dynamic Compression Brace for Pectus Carinatum: Intermediate Results in 286 Patients. Ann Thorac Surg. 2017 Jun;103(6):1742-1749. doi: 10.1016/j.athoracsur.2016.12.019. Epub 2017 Mar 6. PMID 28274516
- [Background] Lee RT, Moorman S, Schneider M, Sigalet DL. Bracing is an effective therapy for pectus carinatum: interim results. J Pediatr Surg. 2013 Jan;48(1):184-90. doi: 10.1016/j.jpedsurg.2012.10.037. PMID 23331813
- [Background] Kang DY, Jung J, Chung S, Cho J, Lee S. Factors affecting patient compliance with compressive brace therapy for pectus carinatum. Interact Cardiovasc Thorac Surg. 2014 Dec;19(6):900-3. doi: 10.1093/icvts/ivu280. Epub 2014 Aug 27. PMID 25164133
- [Background] http://www0.sun.ac.za/ortho/webct-ortho/age/risser.html -].